CLINICAL TRIAL: NCT03995758
Title: MOSES Lithotripsy Technology Applied to Stone Fragmentation During Ureteroscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Original study PI departed the institution
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Marcelino Rivera, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1901990102
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Kidney Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: The patients will be randomized 1:1 to either standard laser lithotripsy or MOSES laser lithotripsy.
Who Masked: Investigator
Masking Description: Surgeons will not be aware of the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard laser lithotripsy (Active Comparator): standard of care for stone fragmentation in ureteroscopy
  Interventions: Device: MOSES
- MOSES laser lithotripsy (Active Comparator): MOSES technology used for stone fragmentation in ureteroscopy
  Interventions: Device: MOSES

INTERVENTIONS:
Device: MOSES — software based modulation of the laser energy delivered from the homium laser source. The software changes the pulsed laser to have two peaks of energy - one to displace water in front of the stone and a second to deliver the laser energy to the stone

SUMMARY:
To determine if the effects of MOSES laser modulation technology can improve the safety and efficiency to laser fragmentation resulting in decreased total laser time, reduced potential for injury to the patient, and total OR time and utilization.

DETAILED DESCRIPTION:
MOSES technology was developed by Lumenis Ltd to maximize the lithotripsy potential of high powered lasers. Typically, a holmium laser unit is used to treat kidney a ureteral stones that are too large to remove en block. Laser lithotripsy allows for a large stone to be partitioned into smaller fragments that can be removed with an endoscopic basket device. Holmium technology has existed for more than 20 years, however, low total power (40 watt) and minimal modulations (Joules and Hertz) of the laser energy by the laser units limited the capacity to improve lithotripsy efficiency.

With the advent of high power (120 watt) lasers with 4 laser cores and developments in software to modulate the laser energy, many more options have emerged for laser lithotripsy of kidney and ureteral stones. At Indiana University Health Physicians Urology, the laser units used for nephrolithotripsy are engineered and produced by Lumenis Ltd. These units are fitted with MOSES technology. Standard laser lithotripsy or MOSES laser lithotripsy can be performed using the same unit and during the same case by simple turning MOSES on or off on the laser touch screen (image 1). MOSES is propriety technology that is software based modulation of the laser energy delivered from the holmium::yag laser source. The software changes the pulsed laser to have two peaks of energy - one to displace the water in front of the stone and the second to deliver the laser energy to the stone. Holmium laser energy dissipates quickly in water, so the displacement of water in front of the stone means more energy is delivered to the stone. With more energy delivery, stone fragmentation is expected to occur more rapidly.

When treating kidney or ureteral stones, there are two distinct surgical approaches. One technique is to use laser lithotripsy to break a stone into tiny pieces called dusting. Dusting technique attempts to turn a stone into a slurry of 2mm or less stone fragments that the patient can pass spontaneously. There are some urologist who promote the use of MOSES technology to improve the efficiency of the dusting technique and reduce operative time. Another approach to endoscopic stone surgery is to laser the stone into fragments to remove with a basket. There is far less laser energy used in this process, however, hard stones and larger stones can take time to fragment. Based on the dusting ureteroscopy data, MOSES technology could still improve fragmentation efficiency and reduce overall operative time.

This is a blinded study. The research coordinator will present to the OR prior to the surgeon to meet with OR staff. At this time, the coordinator will inform the OR staff which group the participant has been randomly assigned. OR staff will be educated to set the laser as instructed by the surgeon but not share whether the MOSES laser lithotripsy is being used. Surgeons will not be aware of the group assignment. The surgeons are only able to adjust the laser energy settings between 0.4-1.0 joules and 4-15 hertz. To control for stone fragment size, surgeons will have to use an 13 french ureteral access sheath independent of ureteral diameter. The MOSES setting is turned on with a touch pad attached to the laser unit. Once the surgeon is ready to laser fragment the stone, the laser will be activated and with the surgeon provided laser energy settings. The laser technician/nurse will follow randomization and add or remove the MOSES option. The surgeons will not be informed if using standard laser or MOSES augmented laser technology. At the conclusion of laser fragmentation, stone basket extraction will occur and once all fragments are removed, the patient will have a ureteral stent placed, awoken, extubated and transferred to the post anesthesia recovery unit. Objective data about laser settings, utilization time and total energy will be obtained at the conclusion of the case. Additionally, the circulating team will record the total OR time. Other variables of interest include blood loss, blood transfusion requirements and complications (utilizing Clavien-Dindo classification) with an expected rate of approximately 1-2%. Subjective grading of stone movement during laser fragmentation as well as stone migration will be recorded.

In addition to the intraoperative variables mentioned above, clinical information including stone size, location, and stone analysis will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Kidney or ureteral stone requiring laser lithotripsy fragmentation

Exclusion Criteria:

* < 18 years of age
* Infectious, struvite stones.
* Atypical collecting system anatomy that prolongs the case (ureteral stricture, malrotated kidney, infundibular stenosis, ureteral duplication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health Physicians Urology, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this study started in June 2019 and concluded in March 2021. Patients for the study were recruited in clinic.
Pre-assignment Details: There are no significant events that occurred after participant enrollment.
Groups:
- Standard Laser Lithotripsy: Standard of care for stone fragmentation in ureteroscopy MOSES: software based modulation of the laser energy delivered from the holmium laser source. The software changes the pulsed laser to have two peaks of energy - one to displace water in front of the stone and a second to deliver the laser energy to the stone
- MOSES Laser Lithotripsy: MOSES technology used for stone fragmentation in ureteroscopy MOSES: software based modulation of the laser energy delivered from the holmium laser source. The software changes the pulsed laser to have two peaks of energy - one to displace water in front of the stone and a second to deliver the laser energy to the stone
Period: Overall Study
Arm/Group | Standard Laser Lithotripsy | MOSES Laser Lithotripsy
Started | 58 | 58
Completed | 58 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Laser Lithotripsy | MOSES Laser Lithotripsy | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 31 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 15 | 16 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of Interest Will be Reduction in Mean Total OR Time
Description: To determine the effects of MOSES laser modulation technology can improve the safety and efficiency to laser fragmentation resulting in decreased total laser time, reduced potential for injury to the patient, and total OR time and utilization.
Time Frame: Postoperative day 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Standard Laser Lithotripsy | MOSES Laser Lithotripsy
Number analyzed (Participants) | 32 | 31
Minutes | 68.2 (35.0) | 64.2 (33.4)

2. Secondary Outcome: Number of Participants With Complications
Description: Clavien Classification of Surgical Complications:
  Grade I: Any deviation from the normal post-operative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions.
  Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgesics, diuretics, electrolytes, and physiotherapy. This grade also includes wound infections opened at bedside.
  Grade II: Requiring pharmacological treatment with drugs other than such allowed for Grade I complications. Blood transfusions and total parenteral nutrition are also included.
  Grade III: Requiring surgical, endoscopic or radiological intervention. Grade IIIa: Intervention not under general anesthesia Grade IIIb: Intervention under general anesthesia Grade IV: Life-threatening complication (including CNS complications) requiring IC/ICU management.
  Grade IVa: Single organ dysfunction (including dialysis) Grade IVb: Multi-organ dysfunction Grade V: Death of a patient
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Laser Lithotripsy | MOSES Laser Lithotripsy
Number analyzed (Participants) | 32 | 31
Participants | 0 | 1

3. Post Hoc Outcome: The Primary Endpoint of Interest Will be Reduction in Mean Total Laser Time
Description: as for outcome 1
Time Frame: Postoperative day 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Standard Laser Lithotripsy | MOSES Laser Lithotripsy
Number analyzed (Participants) | 32 | 31
Seconds | 77.6 (68.3) | 84.5 (107.3)

ADVERSE EVENTS:
Time Frame: The adverse event data was collected for 30 days
Description: Adverse event was collected through surveys
Arm/Group | Standard Laser Lithotripsy | MOSES Laser Lithotripsy
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT03995758/Prot_000.pdf
  • Informed Consent Form (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT03995758/ICF_001.pdf